CLINICAL TRIAL: NCT04060368
Title: STudy to Evaluate the Efficacy and Safety of Endoscopic Sleeve Gastroplasty (ESG) Versus LAparoscopic Sleeve Gastrectomy (LSG) in Obese Subjects With Non-Alcoholic SteatoHepatitis (NASH)
Brief Title: Efficacy and Safety of Endoscopic Sleeve Gastroplasty Versus Laparoscopic Sleeve Gastrectomy in Obese Subjects With NASH
Acronym: TESLA-NASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, UECV, Dr. Javier Crespo, Instituto de Investigación Marqués de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TESLA-NASH
Record Dates: First submitted 2019-07-18; First posted 2019-08-19 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Non-alcoholic Steatohepatitis (NASH)
Keywords: NASH; Obesity; Endoscopic Sleeve Gastroplasty; Laparoscopic Sleeve Gastrectomy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Intervention Model Description: Experimental: Endoscopic Sleeve Gastroplasty with OverStitch® system + Lifestyle modifications Comparator: Laparoscopic Sleeve Gastrectomy + Lifestyle modifications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESG Stitch® system + Lifestyle modifications (Experimental): Endoscopic technique defined as a gastric restriction by means of continuous sutures of the entire gastric wall of the antrum and body, transmurally, in order to simulate a gastric sleeve, in the same way as sleeve gastrectomy surgery. Gastroplasty is performed using an endoscopic suture system (OverStitch, Apollo Endosurgery Inc., Austin, Texas, USA) inserted into a dual-channel endoscope (GIF-2T160, Olympus Medical Systems Corp., Tokyo, Japan).
  Interventions: Procedure: Endoscopic Sleeve Gastroplasty (ESG) with OverStitch® system + Lifestyle modifications
- LSG + Lifestyle modifications (Active Comparator): Minimally invasive surgical technique defined as a gastric restriction by means of an excision approximately 80% of the stomach along the greater curvature.
  Interventions: Procedure: Laparoscopic Sleeve Gastrectomy (LSG) + Lifestyle modifications

INTERVENTIONS:
Procedure: Endoscopic Sleeve Gastroplasty (ESG) with OverStitch® system + Lifestyle modifications — Endoscopic technique defined as a gastric restriction by means of continuous sutures of the entire gastric wall of the antrum and body, transmurally, in order to simulate a gastric sleeve, in the same way as sleeve gastrectomy surgery. Gastroplasty is performed using an endoscopic suture system (OverStitch, Apollo Endosurgery Inc., Austin, Texas, USA) inserted into a dual-channel endoscope (GIF-2T160, Olympus Medical Systems Corp., Tokyo, Japan).
  Arms: ESG Stitch® system + Lifestyle modifications
Procedure: Laparoscopic Sleeve Gastrectomy (LSG) + Lifestyle modifications — Minimally invasive surgical technique defined as a gastric restriction by means of an excision approximately 80% of the stomach along the greater curvature.
  Arms: LSG + Lifestyle modifications

SUMMARY:
The primary objectives of this study are to evaluate the effect of ESG with OverStitch® system (Apollo Endosurgery, Austin, TX, USA) compared to LSG on 1) histological improvement in NASH; 2) all-cause mortality and liver-related outcomes In obese subjects with non-alcoholic steatohepatitis (NASH).

Condition or disease: Non-alcoholic steatohepatitis (NASH) with or without fibrosis Intervention/treatment: ESG with OverStitch® system vs LSG

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 60 years (inclusive) at first screening visit.
2. Must provide signed written informed consent and agree to comply with the study protocol.
3. BMI between 35 and 45 kg/m2 with or without metabolic risk factors (type 2 diabetes, arterial hypertension, dyslipidaemia), and BMI between 30 and 34,9 kg/m2 with type 2 diabetes.
4. Histological confirmation of steatohepatitis in a diagnostic liver biopsy (biopsy obtained in the 6 months prior to randomization or during the selection period) with at least a score of 1 in each component of the NAS score (steatosis with a score of 0 to 3, degeneration by ballooning with a score of 0 to 2 and lobular inflammation with a score of 0 to 3) and:

   * NAS score ≥ 4
   * fibrosis < 4 according to the staging system of CRN fibrosis on NASH
5. For patients with fibrosis ≤ 1, must be associated at least one of the following conditions: metabolic syndrome (NCEP ATP III definition), type 2 diabetes, HOMA-IR >6
6. Absence of other well documented causes of chronic liver disease (alcoholic liver disease, viral hepatitis, cholestasis, autoimmune hepatitis, Wilson's disease, hemochromatosis, alpha 1 antitrypsin deficiency)
7. Patients agree to have 1 liver biopsy after 96 weeks after intervention

Exclusion Criteria:

1. Known heart failure (Grade I to IV of the classification of the New York Heart Association).
2. History of efficient bariatric surgery within 10 years prior to Screening.
3. Patients with a history of clinically significant acute cardiac event in the 6 months prior to selection, such as: acute cardiovascular event, cerebrovascular accident, transient ischemic attack, or coronary heart disease (angina pectoris, myocardial infarction, revascularization procedures).
4. Weight loss of more than 5% in the 6 months prior to randomization.
5. Recent or current background of significant consumption of alcoholic beverages (<5 years). In the case of men, significant consumption is usually defined as more than 30 g of pure alcohol per day. In the case of women, it is usually defined as more than 20 g of pure alcohol per day.
6. Liver cirrhosis.
7. Non-cirrhotic portal hypertension.
8. Esophagogastric varices.
9. Hepatocellular carcinoma
10. Portal thrombosis.
11. Pregnancy.
12. Refusal to give informed consent.
13. Any medical condition that could reduce life expectancy to less than 2 years, including known cancers.
14. Signs of any other unstable or clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, neoplastic or psychiatric disease without treatment.
15. Instability or mental incompetence, so that the validity of the informed consent or the ability to comply with the study are uncertain.
16. Antibodies positive for the human immunodeficiency virus.
17. Descompensated liver disease with the following hematologic and biochemical criteria:

    * Aspartate aminotransferase (AST) and / or ALT> 10 x upper limit of normal (ULN)
    * Total bilirubin> 25 μmol / l (1.5 mg / dl)
    * Standardized international index> 1.4
    * Platelet count <100 000 / mm3
18. Serum creatinine levels> 135 μmol / l (> 1.53 mg / dl) in men and> 110 μmol / l (> 1.24 mg / dl) in women.
19. Significant renal disease, including nephritic syndrome, chronic kidney disease (patients with markers of hepatic injury or estimated glomerular filtration rate [eGFR] of less than 60 ml / min / 1.73 m2). If an abnormal value is obtained at the first screening visit, the eGFR measurement may be repeated before randomization within the following time frame: minimum 4 weeks after the initial test and maximum 2 weeks before the expected randomization. An abnormal repeated eGFR (less than 60 ml / min / 1.73 m2) leads to exclusion from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects undergoing ESG relative to LSG achieving resolution of NASH without worsening of fibrosis | Measurement at 96 weeks
  To evaluate the effect of ESG compared to LSG on liver histology in obese subjects with NASH with or without fibrosis by assessing the following endpoint: The proportion of subjects undergoing ESG relative to LSG achieving NASH resolution without worsening of fibrosis. NASH resolution is defined as the disappearance of ballooning and the disappearance or persistence of minimal lobular inflammation (grade 0 or 1) The worsening of fibrosis is defined as the progression of at least one stage.
Proportion of subjects undergoing ESG relative to LSG with cardiovascular and liver-related death events | Measurement at 96 weeks
  To evaluate the effect of ESG compared to LSG on liver histology in obese subjects with NASH with fibrosis by assessing the following endpoint: The proportion of subjects undergoing ESG relative to LSG achieving improvement of liver fibrosis of at least one stage.

SECONDARY OUTCOMES:
Proportion of subjects undergoing ESG relative to LSG achieving improvement in liver histology according to the NASH-CRN scoring | Measurement at 96 weeks
  Percentage of patients with at least 1 point improvement
Changes in the liver enzymes | Measurement at 96 weeks
  ALT, AST, GGT, AP (U/L)
Changes in lipid parameter | Measurement at 96 weeks
  Cholesterol, LDL, HDL, Triglycerides (mg/dL)
Changes in noninvasive markers of fibrosis and steatosis | Measurement at 96 weeks
  Fatty Liver Index (FLI) (<30; 30-60; >60)
Changes in noninvasive markers of fibrosis and steatosis | Measurement at 96 weeks
  Hepatic steatosis index (HSI) (<30; 30-36; >36)
Changes in noninvasive markers of fibrosis and steatosis | Measurement at 96 weeks
  NAFLD fibrosis score (NFS) (<-1.455; -1.455-0.676; >0.676)
Changes in noninvasive markers of fibrosis and steatosis | Measurement at 96 weeks
  AST to Plateler ratio index (APRI) (<1, >1)
Changes in noninvasive markers of fibrosis and steatosis | Measurement at 96 weeks
  Fibrosis-4 (FIB-4) (<1.30; 1.30-2.67; >2.67)
Changes in noninvasive markers of fibrosis and steatosis | Measurement at 96 weeks
  Hepamet fibrosis score (HFS) (<0.12; 0.12-0.47; >0.47)
Changes in body weight | Measurement at 96 weeks
  body weight
Changes in inflammatory markers | Measurement at 96 weeks
  Ferritin in ng/mL
Changes in inflammatory markers | Measurement at 96 weeks
  C-rective protein (CRP) in mg/dL
Changes in inflammatory markers | Measurement at 96 weeks
  High sensitivity C-reactive protein (hs-CRP) in mg/L
Changes in inflammatory markers | Measurement at 96 weeks
  Interleukin 6 (IL-6) in pg/mL
Changes in inflammatory markers | Measurement at 96 weeks
  Interleukin 1 beta (IL-1b) in pg/mL
Changes in inflammatory markers | Measurement at 96 weeks
  Tumor necrosis factor alpha (TNFa) in pg/mL
Changes in serum expression of incretins | Measurement at 96 weeks
  serum expression of incretins
Changes in mineral metabolism parameters. | Measurement at 96 weeks
  Parathormone (PTH) (pg/mL), 25(OH)D (ng/mL), PINP, b-CTX (ng/mL)
Changes in gut microbiota | Measurement at 96 weeks
  Analysis using 16S rRNA sequencing from stool samples
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Glucose in mg/dL
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Hemoglobin A1c (HbA1c) in %
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Homeostatic model assessment for insulin resistance (HOMA-IR) (not unit)
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Adponectin in ug/mL
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Retinol binding protein 4 (RBP-4) in ug/mL
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Monocyte chemoattractant protein-1 (MCP-1) in ug/mL
Changes in glucose homeostasis markers and insulin resistance | Measurement at 96 weeks
  Plaminogen activator inhibitor-1 (PAI-1) in ug/mL
Incidence of adverse events | Measurement at 96 weeks
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Hospitl Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

REFERENCES:
- [Result] Cuadrado A, Orive A, Garcia-Suarez C, Dominguez A, Fernandez-Escalante JC, Crespo J, Pons-Romero F. Non-alcoholic steatohepatitis (NASH) and hepatocellular carcinoma. Obes Surg. 2005 Mar;15(3):442-6. doi: 10.1381/0960892053576596. PMID 15826485
- [Result] Singh S, Allen AM, Wang Z, Prokop LJ, Murad MH, Loomba R. Fibrosis progression in nonalcoholic fatty liver vs nonalcoholic steatohepatitis: a systematic review and meta-analysis of paired-biopsy studies. Clin Gastroenterol Hepatol. 2015 Apr;13(4):643-54.e1-9; quiz e39-40. doi: 10.1016/j.cgh.2014.04.014. Epub 2014 Apr 24. PMID 24768810
- [Result] Pais R, Charlotte F, Fedchuk L, Bedossa P, Lebray P, Poynard T, Ratziu V; LIDO Study Group. A systematic review of follow-up biopsies reveals disease progression in patients with non-alcoholic fatty liver. J Hepatol. 2013 Sep;59(3):550-6. doi: 10.1016/j.jhep.2013.04.027. Epub 2013 May 9. PMID 23665288
- [Result] Vernon G, Baranova A, Younossi ZM. Systematic review: the epidemiology and natural history of non-alcoholic fatty liver disease and non-alcoholic steatohepatitis in adults. Aliment Pharmacol Ther. 2011 Aug;34(3):274-85. doi: 10.1111/j.1365-2036.2011.04724.x. Epub 2011 May 30. PMID 21623852
- [Result] Machado M, Marques-Vidal P, Cortez-Pinto H. Hepatic histology in obese patients undergoing bariatric surgery. J Hepatol. 2006 Oct;45(4):600-6. doi: 10.1016/j.jhep.2006.06.013. Epub 2006 Jul 25. PMID 16899321
- [Result] Boza C, Riquelme A, Ibanez L, Duarte I, Norero E, Viviani P, Soza A, Fernandez JI, Raddatz A, Guzman S, Arrese M. Predictors of nonalcoholic steatohepatitis (NASH) in obese patients undergoing gastric bypass. Obes Surg. 2005 Sep;15(8):1148-53. doi: 10.1381/0960892055002347. PMID 16197788
- [Derived] Lavin-Alconero L, Fernandez-Lanas T, Iruzubieta-Coz P, Arias-Loste MT, Rodriguez-Duque JC, Rivas C, Cagigal ML, Montalban C, Useros AL, Alvarez-Cancelo A, Garcia-Saiz M, Crespo-Garcia J. Efficacy and safety of endoscopic sleeve gastroplasty versus laparoscopic sleeve gastrectomy in obese subjects with Non-Alcoholic SteatoHepatitis (NASH): study protocol for a randomized controlled trial (TESLA-NASH study). Trials. 2021 Oct 30;22(1):756. doi: 10.1186/s13063-021-05695-7. PMID 34717726